CLINICAL TRIAL: NCT02677103
Title: Comparison of the Effect of Radial Shock Wave, Ultrasound-guided Needle Puncture, and Combination of Both in the Treatment of Calcific Tendinitis of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120801R
Record Dates: First submitted 2014-09-02; First posted 2016-02-09 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Calcific Tendinitis of the Shoulder
Keywords: Radial shock wave therapy,calcific tendinitis, ultrasound guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RSWT group (Experimental): The RSWT was delivered at 2 Hz with 2000 shock waves and the energy level of 0.26mJ/mm2 in calcific tendinitis of shoulder. RSWT will be performed once per week, and will be continued for 3 weeks.
  Interventions: Device: radial extracorporeal shock wave therapy
- USNP group (Experimental): All needle punctures will be guided by ultrasound (US). The puncture needle is a 3.8cm 22# needle attached on a 5ml syringe. Before puncture, the skin of the puncture site will be sterilized with better iodine, and the transducer will be covered with a sterilized plastic bag. After injecting 3cc 1% Xylocain in the subcutaneous tissue, muscle layer and subdeltoid bursa, multiple back-and-forth puncture about 10-20 times (depending on the size of the plaques) within the calcific plaques will be performed. The needle tract will be monitored by ultrasound to make sure the needle penetrated through the calcific plaque, but does not penetrate the rotator cuff.
  Interventions: Procedure: ultrasound-guided needle puncture
- RSWT plus USNP (Experimental): In this group, each subject will receive radial shock wave therapy after ultrasound-guided needle puncture, as described in the previous paragraphs
  Interventions: Procedure: RSWT and USNP

INTERVENTIONS:
Device: radial extracorporeal shock wave therapy — he RSWT was delivered at 2 Hz with 2000 shock waves and the energy level of 0.26mJ/mm2 in calcific tendinitis of shoulder.
  Other Names: RSWT
  Arms: RSWT group
Procedure: ultrasound-guided needle puncture — After injecting 3cc 1% Xylocain in the subcutaneous tissue, muscle layer and subdeltoid bursa, multiple back-and-forth puncture about 10-20 times (depending on the size of the plaques) within the calcific plaques will be performed.
  Other Names: USNP
  Arms: USNP group
Procedure: RSWT and USNP — each subject will receive radial shock wave therapy after ultrasound-guided needle puncture, as described in the previous paragraphs.
  Arms: RSWT plus USNP

SUMMARY:
Calcific tendinitis of the shoulder is a common enthesopathy, and is characterized by inflammation around calcium hydroxyapatite crystal deposits, usually located in the supraspinatus tendon, near its insertion place.1 The disease mainly affects individuals between 30 and 50 years of age, is painful in 50% of patients and frequently leads to considerable restriction of motion.2,3 It goes through three distinct stages: a precalcific stage (metaplasia of matrix), calcific stage (calcification of matrix and resorption of calific deposits), and a postcalcific stage (reconstitution of matrix).

Classifications of calcific tendinitis have been proposed previously. Gartner proposed a classification based on plain films of the shoulder: type I deposits were sharply outlined and densely structured. Type III deposits had a cloudy outline and were transparent in structure. Type II deposits were features of both.4 Type III plaques have a tendency to resorb. Due to the progress of musculoskeletal ultrasound over the past decade, classification of the calcific tendinitis based on ultrasound findings was also proposed: arc-shaped (an echogenic arc with clear shadowing), fragmented or punctate (at least 2 separated echogenic spots or plaques with or without shadowing), nodular (an echogenic nodule without shadowing), and cystic (a bold echogenic wall with an anechoic area).5 Plaques that appear fragmented, nodular, or cystic on ultrasound are considered in the resorptive phase.

The treatment of patients with calcific tendinitis is typically conservative. The reported success rates vary between 30 and 85%.6 If the pain becomes chronic or intermittent after several months of conservative treatment, arthroscopic and open procedures are available to curette the calcium deposit, and additional subacromial decompression can be performed if necessary.7,8 As an alternative, minimally invasive extracorporeal shock wave therapy (ESWT) has been postulated to be an effective treatment option for treating calcific tendinopathy of the shoulder, before surgery.9-12 In recent years, radial shock wave has been developed. A radial shock wave is a low- to medium-energy shock wave that is pneumatically generated through acceleration of a projectile inside the handpiece of the treatment device and then transmitted radially from the tip of the applicator to the target zone. Radial shock wave showed a low pressure and a considerably longer rise time than extracorporeal shock wave. In radial shock wave therapy (RSWT), the focal point is not concentrated on the target zone, as occurred in ESWT, but on the tip of applicator. 13 Another new method of conservative treatment of calcific tendinopathy is ultrasound-guided fine-needle repeated puncture of the calcific plaque, as shown in previous study.14,15 The new method has the advantage of being easily operative, cheap, safe, and has a proven high success rate. Although percutaneous needle aspiration with a large size needle(≥ 18# needle) alleviates symptoms in up to 60% of patients and resolves the deposits in 40% to 74%,16,17 the larger size needle could result in tendon injury.

In clinical practice, combination of radial shock wave therapy and ultrasound-guided fine needle repeated puncture is frequently used and shows promising results, however, scientific report has been rarely published before.18 The purpose of this study is to compare the efficacy of RSWT, ultrasound-guided fine needle puncture (USNP), and combination of RSWT and USNP in the treatment of calcific tendinitis of shoulder.

DETAILED DESCRIPTION:
A prospective, randomized, controlled trial will be conducted.Thirty patients in each group with calcific tendinitis of shoulder from the outpatient clinic of Department of Physical Medicine and Rehabilitation in Shin Kong Wu Ho-Su Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20~75 y
2. Subject with calcific tendinitis of the shoulder.
3. Fulfill inclusion criteria and not meet exclusion criteria.

Exclusion Criteria:

pregnancy, clotting disorders, anticoagulant or antiplatelet treatment, cardiac pacemaker, chronic inflammatory joint disease, infections or tumors of the shoulder, adhesive capsulitis, hyperalgia of the shoulder due to resorption of a calcific deposit, and calcification of type III as defined by Gartner or nodular or cystic type of calcification defined by Chiou.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | 1.5 month, 3 months after the treatment.
  VAS; horizontal lines of 100 mm, with 0 indicating no pain on the left and 100 indicating very severe pain on the right.
  A VAS has been found to be reliable and sensitive tool for measuring pain, with test-retest reliability of >0.90. In previous studies of subjects treated for various shoulder disorders, the responsiveness of VAS for pain was moderate to good.

SECONDARY OUTCOMES:
Active ROM and passive ROM | .5 month, 3 months after the treatment.
  conventional goniometer in accordance with the guideline of the American Academy of the Orthopedic Surgeons19 and included abduction in the frontal plane, forward flexion, and internal rotation and external rotation with the arm in 0 degrees of abduction
General health status: 36-Item Shot-Form Health Survey (SF-36) | 1.5 month, 3 months after the treatment.
  The SF-36, the psychometric properties of which have been established for the Chinese language, is a generic measure of quality of life comprising 8 subscales for physical functioning, social functioning, role limitations (physical problems), role limitations (emotional problems), mental health, vitality, pain, and general health perception. Each subscale generates a score from 0 to 100, with higher score indicating better health. From these 8 health concepts, 2 summary scales, for physical health and mental health, can be computed.
Shoulder problems | .5 month, 3 months after the treatment.
  Shoulder problems will be measured by means of Constant Score, which is a 100-point score system that included 15 points for pain, 20 points for activities of daily living, 40 points for shoulder motion, and 25 points for the muscle power of the affected arm.
Patients' satisfaction | 1.5 month, 3 months after the treatment.
  Patients' satisfaction will be classified as very satisfactory, satisfactory, partially satisfactory, and unsatisfactory, scoring 1, 2, 3, and 4 points, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan